CLINICAL TRIAL: NCT02937727
Title: Evaluate the Safety and Effectiveness of 3T MRI Compatible and Long-term LFP Recordable Deep Brain Stimulation on PD Patients
Brief Title: MRI Compatible and Long-term LFP Recordable Deep Brain Stimulation on PD Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINS-021
Record Dates: First submitted 2016-10-13; First posted 2016-10-19 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2016-10

CONDITIONS: Idiopathic Parkinson Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI compatible and LFP recordable implantable stimulator (Experimental)
  Interventions: Device: 3T MRI compatible and LFP recordable G106R of Beijing Pins medical.

INTERVENTIONS:
Device: 3T MRI compatible and LFP recordable G106R of Beijing Pins medical.

SUMMARY:
Deep Brain Stimulation represents the golden standard for surgical treatment of Parkinson's disease (PD), but it is not optimally effective for controlling every motor sign and adverse events are not so infrequent. Therefore,other approaches should be considered. New Approaches in MRI at 3T and long-term local field potential (LFP) recording are very important to target subthalamic nucleus (STN) and understand mechanisms of DBS on Parkinson Patients. This study aims at evaluating the safety and effectiveness of 3T MRI Compatible and LFP recordable deep brain stimulation on PD patients. The Chronically LFP recording using G106R is for two goals: 1) Evaluate the performance of long-term recordable neural simulation. 2) Study long-term clinical and electrophysiology effects of deep brain stimulation on STN.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18，≤75，idiopathic Parkinson's disease，both male and female
2. MMSE score ≥24
3. H-Y score ≥2.0 on the medicine off situation
4. UPDRS-III score≥30 on the medicine off situation
5. The duration of this disease ≥5 years
6. Ability to provide informed consent as determined by preoperative neuropsychological assessment
7. History of appropriate response to dopaminergic medication, with at least a 30% improvement in motor UPDRS with L-DOPA by history or in-clinic testing, for the PD patients
8. Excellent responsiveness to levodopa
9. ≥6h in medicine off state

Exclusion Criteria:

1. Lack of ability to provide informed consent as determined by preoperative neuropsychological assessment
2. Otherwise not eligible for DBS surgery, for example known inability to undergo anesthesia
3. Hydrocephalus，brain atrophy，cerebral infarction ，cerebralvascular diseases
4. Patients who are unable to follow verbal instructions
5. Other severe pathological chronic condition that might confound treatment effects or interpretation of the data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
UPDRS part III | 1 month,3 months, 6 months and 12months
Local Field Potential Recordings using G106R | 1 month,3 months, 6 months and 12months

SECONDARY OUTCOMES:
UPDRS part III | 1, 3 months of stimulation
UPDRS part II | 1, 3 months stimulation
Levodopa Equivalent Dose | 1, 3 months stimulation
  Drug Therapy are definied as levodopa equivalent dose,which is devodopa containing or dopamine agonist containing medications
Local Field Potential Recordings using G106R | 1 month, 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Qilu Hospital of Shandong University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhang G, Yu H, Chen Y, Gong C, Hao H, Guo Y, Xu S, Zhang Y, Yuan X, Yin G, Zhang JG, Tan H, Li L. Neurophysiological features of STN LFP underlying sleep fragmentation in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2024 Nov 18;95(12):1112-1122. doi: 10.1136/jnnp-2023-331979. PMID 38724231